CLINICAL TRIAL: NCT01321528
Title: Pilot Clinical Trial of Inquiry-based Stress Reduction (IBSR) Program for Health Care Professionals
Brief Title: Trial of Inquiry-based Stress Reduction (IBSR) Program for Health Care Professionals
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Yaffa Lerman MD, Tel Aviv Sourasky Medical Center
Other Study IDs: TASMC 11 YL 0037 CTIL
Record Dates: First submitted 2011-03-10; First posted 2011-03-23 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Behavioral Symptoms
MeSH Terms: conditions — Behavioral Symptoms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IBSR Intervention group: 30 nurses in the geriatric departments in TASMC

SUMMARY:
The IBSR (Inquiry-based stress reduction) intervention, developed by Byron Katie (www.thework.com), trains subjects to reduce their perceived level of stress by self-inquiry of their thoughts and beliefs connected to stressful circumstances or symptoms. This meditative process, named "The Work", enables the participants to identify and question the stressful thoughts that cause their suffering. The core of IBSR is simply four questions and a turnaround, which is a way of experiencing the opposite of what the participant believes. This process is simple, powerful and can be easily implemented in daily life.

Therefore, on the basis of previous data and beneficial observations the investigators postulate that the clinical utility of IBSR mediation program may alleviate stress and rate of burnout and improve quality of life among health care professionals. Thus, we will conduct a pilot/feasibility Observational study designed to:

* Assess feasibility of a IBSR intervention by examining attendance, drop-out rates, and program satisfaction.
* investigate whether IBSR intervention is efficacious in alleviating stress and rate of burnout and improving quality of life among health care professionals.

DETAILED DESCRIPTION:
Study Goals To investigate whether IBSR intervention is efficacious in alleviating stress and rate of burnout and improving quality of life among health care professionals.

Study methodology The proposed study is pilot/feasibility intervention study with pre and post measures. 30 participants will receive Inquiry-based stress reduction (IBSR) group intervention.

Population The pilot intervention group will consist 30 nurses at the Geriatric Rehabilitation Department in the Tel Aviv Sourasky Medical Center (TASMC) who are willing to participate in this study.

Data collection procedures

1. Assessments will be taken at an initial baseline orientation and at the end of the 12-week intervention.
2. One week before IBSR classes will start, a baseline orientation will be held at this session, informed consent will be obtained, baseline data will be collected, and a brief overview of the IBSR program will be provided, which will highlight the 12-week class schedule.

Intervention

1. Subjects will receive weekly 3.5 hour sessions conducted by two facilitators trained in IBSR and certified by BKI to conduct this intervention.
2. Class size will range from 12-16 participants.
3. All the sessions will be standardized and follow the training manual developed to maintain consistency in the program.
4. Subjects will receive a training manual and CD's to support home practice of various forms of inquiry practices.
5. The training manual will include weekly exercises, and program content related to the content identified below. In addition, the manual will include a weekly diary for recording homework practice activities.

The IBSR-BC program is a 12-week program adapted for consideration of health professionals well-being. During the process, participants will be encouraged to identify and inquire about their stressful thoughts: regarding health and illness, relationships with others, Beliefs that prevent them to promote their health, self judgments, perception of death and suffering. This intervention provides for management of specific emotional/psychological symptoms (stress, anxiety, depression) and physical symptoms, such as fatigue and sleeps disorders and enables the participants to inquire and be relieved of their stressful thoughts, and emotions caused by these thoughts. Through the use of self-inquiry practices subjects are taught to increase awareness of their thoughts and feelings, to observe their emotional and physical responses during situations perceived by them as stressful, and allow their mind to return to its true, peaceful, creative nature. Through the process of self inquiry, subjects take an active role in investigating their stressful thoughts, and by this regulating their stress and managing symptoms and emotions, thus enabling them to cope better with with emotional stress and burnout.

Throughout the 12-week IBSR (HCP - health care professionals) program, all subjects will be requested to formally meditate and perform self inquiry exercises alone or with a partner for a minimum of 15 min per day.

ELIGIBILITY:
Inclusion Criteria:

1. nurses in the geriatric departments in TASMC
2. Willing to sign an informed consent
3. Age 18-67

Exclusion Criteria:

nursing assistants employees

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 participants nurses in the geriatric departments in TASMC
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yaffa Lerman, MD, Principal Investigator — Tel Aviv Sourasky Medical canter; Shahar Lev Ari, PHD, Study Director — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel